CLINICAL TRIAL: NCT03081390
Title: Mechanisms of Increased Cardiovascular Disease Risk in Women With Migraine
Brief Title: Migraine and CVD Risk in Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 826251
Record Dates: First submitted 2017-02-16; First posted 2017-03-16 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: There are four total groups of participants, stratified according to migraine status (yes/no) and obesity status (yes/no). All undergo the same experimental phenotyping procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No migraine, normal weight (Experimental): * Mixed meal tolerance testing
  * Skin conductance & cold pressor test
  * Flow-mediated dilation testing
  Interventions: Other: Mixed meal tolerance testing; Other: Skin conductance & cold pressor test; Other: Flow-mediated dilation testing
- No migraine, obese (Experimental): * Mixed meal tolerance testing
  * Skin conductance & cold pressor test
  * Flow-mediated dilation testing
  Interventions: Other: Mixed meal tolerance testing; Other: Skin conductance & cold pressor test; Other: Flow-mediated dilation testing
- Migraine, normal weight (Experimental): * Mixed meal tolerance testing
  * Skin conductance & cold pressor test
  * Flow-mediated dilation testing
  Interventions: Other: Mixed meal tolerance testing; Other: Skin conductance & cold pressor test; Other: Flow-mediated dilation testing
- Migraine, obese (Experimental): * Mixed meal tolerance testing
  * Skin conductance & cold pressor test
  * Flow-mediated dilation testing
  Interventions: Other: Mixed meal tolerance testing; Other: Skin conductance & cold pressor test; Other: Flow-mediated dilation testing

INTERVENTIONS:
Other: Mixed meal tolerance testing — An intravenous catheter is placed for serial blood draws for inflammatory markers and ancillary studies. The participant consumes a test meal, and measurements are made for 4 hours.
Other: Skin conductance & cold pressor test — Skin conductance will be monitored continuously with 2 electrodes placed on the plantar surface of the foot. To induce pain, we will use the cold pressor test. Participants submerge one hand in a bath with iced water (2-4ºC) for 2 minutes. Blood pressure and heart rate are monitored every minute starting 5 minutes before the cold pressor test and for 10 minutes after the participant withdraws the hand from the bath. This testing will be performed at baseline and post-meal.
Other: Flow-mediated dilation testing — At baseline and post-meal, we will assess flow-mediated dilation at the brachial artery using well-validated ultrasound techniques.

SUMMARY:
The primary goal of this study is to test the effects of a high-fat, high-carbohydrate mixed meal on candidate modulators of cardiovascular disease risk (inflammation, vascular reactivity, sympathetic nervous system tone, and response to pain) in young adult women with migraine compared with healthy young women. This is study enrolling both cases (women with migraine) and controls (women without migraine), with equal numbers of normal weight and obese women in each group. Participants will undergo a telephone screening and a single day in-person study visit.

ELIGIBILITY:
Inclusion Criteria (all):

* Female 18-35 years of age, inclusive
* BMI 18.5-24.9 kg/m2, inclusive
* BMI ≥30 kg/m2

Inclusion Criteria (cases only):

* Diagnosis of migraine per ICHD-3-beta (1-10 migraine days per month)

Exclusion Criteria (all):

* Smoking (current or former)
* Chronic use of medications, including oral contraceptives
* Major medical or psychiatry illness (e.g. diabetes, fibromyalgia, major depression/anxiety)
* Pregnant or nursing
* Allergies or sensitivity to any of the ingredients of the meal
* Inability to fast for 10 hours and/or abstain from caffeine intake for 24 hours
* Treatment with antibiotics or steroids within the previous 3 months
* Treatment with NSAIDs within the previous 1 week

Exclusion Criteria (controls only):

* Migraine headaches, or headaches other than tension-type headaches with a frequency of 1 or fewer days per month

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-reported female.
Enrollment: 30 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
LPS area under the curve (AUC) | LPS is measured at baseline every 30 minutes for 4 hours.
  The primary study endpoint is lipopolysaccharide (LPS) area under the curve (AUC) during MMTT.

SECONDARY OUTCOMES:
Flow-mediated dilation (FMD) | FMD is measured at baseline and 2.5 hours after MMTT.
  Vascular reactivity via brachial artery ultrasound, expressed as flow-mediated dilation (% of baseline diameter, normalized).
Sympathetic tone at rest and with painful stimulus | Sympathetic tone at rest and with painful stimulus are measured at baseline and 3 hours after MMTT.
  Sympathetic tone via skin conductance is expressed as mean skin conductance level (SCL) in microsiemens, and assessed at rest and following a pain stimulus (cold pressor test).

CONTACTS AND LOCATIONS:
Overall Officials: Shana E McCormack, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
After the primary publication is complete, interested investigators can request these data without identifiers. The study team will evaluate the request for scientific rigor and ensure consistency with our protocol, and then provide data without identifiers via secure file-share. This will include the subset of participants who indicated their data could be used for ancillary and/or future studies.